CLINICAL TRIAL: NCT07253168
Title: Intratumoral Microbiota in Breast Cancer: A Prospective Discovery Study Integrating Tumor/Adjacent Normal Tissue, Estrobolome, and Gut Microbiota Analyses, With Stratification by Molecular Subtypes
Brief Title: Tumor Integrating Gut Microbiota in bREast Cancer
Acronym: TIGER-BC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 8051
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing surgery for breast cancer (Experimental): single-arm discovery study with consecutive enrollment of eligible patients undergoing surgery for primary breast cancer
  Interventions: Procedure: Surgery for breast cancer

INTERVENTIONS:
Procedure: Surgery for breast cancer — To investigate the intratumoral microbiota in breast cancer and integrate these findings with gut microbiota analyses, including estrobolome characterization, to explore potential microbial-host interactions influencing tumor biology across molecular subtypes
  Other Names: Characterization of intratumoral microbiota

SUMMARY:
Study on patients undergoing surgery for breast cancer. Objective: to characterize the intratumoral microbiota and integrate these findings with clinicopathologic data, the estrobolome, and gut microbiota, with analyses stratified by molecular subtype (Luminal A, Luminal B, HER2-enriched [human epidermal growth factor receptor 2-enriched], and TNBC [triple-negative breast cancer]).

Enrollment: consecutive recruitment in the operating room based on the availability of biopsy/histological material.

Samples: tumor tissue, adjacent normal tissue; urine (for indirect assessment of estrobolome activity); and stool. Strict anti-contamination measures will be implemented.

Exploratory outcomes: differences across subtypes, associations with features of the TME (tumor microenvironment), including TILs (tumor-infiltrating lymphocytes), and markers of progression or treatment resistance

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years with primary, non-metastatic breast cancer (BC) undergoing surgery.
* Availability of sufficient tumor and adjacent normal tissue for research purposes after completion of diagnostic sampling.
* Written informed consent

Exclusion Criteria:

* Active systemic infection or fever >38.0°C within 72 h pre-surgery.
* Antibiotics within 14 days pre-sampling (recorded; analyses adjusted).
* Prior ipsilateral BC surgery for current lesion (except re-excision with fresh tissue).
* Any condition preventing compliance with the study protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Breast cancer-associated microbial signatures | 12 months
  To characterize intratumoral microbial signatures (composition and inferred function) across breast cancer (BC) molecular subtypes (Luminal A, Luminal B, HER2-enriched, TNBC) using contamination-aware pipelines

SECONDARY OUTCOMES:
Comparison of microbial signatures | 12 months
  To compare microbial signatures between tumor and adjacent normal tissue (paired design)
Association between microbial and host features | 12 months
  To explore associations between intratumoral microbial features and clinicopathologic and host variables

CONTACTS AND LOCATIONS:
Overall Officials: Brunella Posteraro, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS